CLINICAL TRIAL: NCT03761082
Title: Post Marketing Surveillance of PIRESPA® TAB 200mg (Pirfenidone) for Evaluating the Safety and Efficacy
Status: Completed | Type: Observational
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ID-PIR-401
Record Dates: First submitted 2018-08-24; First posted 2018-12-03 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NA(observation study) — NA(observation study)

SUMMARY:
Post-marketing surveillance of Pirfenidone

DETAILED DESCRIPTION:
Pirfenidone (Pirespa®) is an anti fibrotic drug, which was approved in 2012 in the Republic of Korea for the treatment of patients with idiopathic pulmonary fibrosis (IPF). A post-marketing survey was conducted following the approval to obtain data on the safety and efficacy of pirfenidone for IPF treatment in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

* Among patients diagnosed as idiopathic pulmonary fibrosis, only those who have used the testing drug under the general medical conditions for a certain investigation period after the beginning of the investigation and also signed a the "Personal Information Utilization Agreement" form. However, for those who have already received the drug before the beginning of the investigation, only the subjects whose medical record can be used are included.

Exclusion Criteria:

1. Subjects who is hypersensitive to the active ingredient or additives of this drug
2. Subjects who have severe hepatopathy
3. Subjects who have severe renal disorder (creatinine clearance<30mL/min) or a terminal renal disease treated by dialysis
4. Subjects who received a combined treatment of fluvoxamine
5. Subjects who have genetic problems, such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: residents of Korea, in real-world practice
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The change from baseline to week 48 in the percentage of the predicted FVC | up to 48 weeks
  In case of administering this drug for more than 12 weeks after registration in the investigation, response evaluation is conducted every 12 weeks (12,24,36,48 weeks) and records are investigated before administration of this drug and after 12, 24,36,48 weeks of administration.

SECONDARY OUTCOMES:
Incidence of adverse event after this drug administration in general medical | 48 weeks
  Any adverse events occurred after this drug dosing will be recorded. Description of adverse event(s) including type of adverse event(s), onset/end date, severity, action taken, causal relationship to the drug and investigator's view on the adverse event(s) will be captured, whether it is related to the drug or not and until follow up visit more than 1 time during the surveillance period.
  Lab abnormalities and changes in vital signs are considered to be adverse events only if they result in discontinuation from the study, necessitate therapeutic medical intervention, and/or if the investigator considers them to be adverse events.

IPD SHARING:
Plan to Share IPD: Undecided
not yet discussed on the issue

REFERENCES:
- [Derived] Chung MP, Park MS, Oh IJ, Lee HB, Kim YW, Park JS, Uh ST, Kim YS, Jegal Y, Song JW. Safety and Efficacy of Pirfenidone in Advanced Idiopathic Pulmonary Fibrosis: A Nationwide Post-Marketing Surveillance Study in Korean Patients. Adv Ther. 2020 May;37(5):2303-2316. doi: 10.1007/s12325-020-01328-8. Epub 2020 Apr 15. PMID 32297284